CLINICAL TRIAL: NCT04603027
Title: A Phase 2, Multicenter, Randomized, Double-Blind, Placebo-Controlled, Parallel-Cohort, Dose-Ranging Study Investigating the Effect of EDP1815 in the Treatment of Mild to Moderate Plaque Psoriasis
Brief Title: A Phase 2 Study Investigating the Effect of EDP1815 in the Treatment of Mild to Moderate Plaque Psoriasis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Evelo Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: EDP1815-201
Record Dates: First submitted 2020-10-16; First posted 2020-10-26 (Actual); Results first posted 2022-12-19 (Actual); Last update posted 2022-12-19 (Actual); Status verified 2022-09

CONDITIONS: Psoriasis; Plaque Psoriasis
Keywords: PSO; mild psoriasis; moderate psoriasis; plaque psoriasis; psoriasis; EDP1815
MeSH Terms: conditions — Psoriasis

STUDY DESIGN:
Intervention Model Description: This is a multicenter, randomized, double-blind, placebo-controlled, parallel-cohort, dose-ranging study of participants with mild to moderate plaque psoriasis
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Experimental): 75 subjects with mild to moderate psoriasis; 50 on EDP1815, 25 on placebo. Dose = 0.8 x 10^11 cells, capsule, once daily, 16 weeks
  Interventions: Drug: EDP1815; Drug: Placebo
- Cohort 2 (Experimental): 75 subjects with mild to moderate psoriasis; 50 on EDP1815, 25 on placebo. Dose = 3.2 x 10^11 cells, capsule, once daily, 16 weeks
  Interventions: Drug: EDP1815; Drug: Placebo
- Cohort 3 (Experimental): 75 subjects with mild to moderate psoriasis; 50 on EDP1815, 25 on placebo. Dose = 8.0 x 10^11 cells, capsule, once daily, 16 weeks
  Interventions: Drug: EDP1815; Drug: Placebo

INTERVENTIONS:
Drug: EDP1815 — EDP1815 is an orally administered, pharmaceutical preparation of a single strain of bacteria
Drug: Placebo — Placebo oral capsule

SUMMARY:
This Phase 2 study has been designed to investigate the clinical safety and efficacy of EDP1815 and to identify an optimal dose in subjects with mild to moderate psoriasis.

DETAILED DESCRIPTION:
This is a multicenter, randomized, double-blind, placebo-controlled, parallel-cohort, dose-ranging study of participants with mild to moderate plaque psoriasis. This Phase 2 study has been designed to investigate the clinical safety and efficacy of EDP1815 and to identify an optimal dose in subjects with mild to moderate psoriasis.

ELIGIBILITY:
Key Inclusion Criteria:

1. Males or females ≥18 and ≤70 years old at the time of informed consent.
2. A documented diagnosis of plaque psoriasis for ≥6 months.
3. Have mild to moderate plaque psoriasis with plaque covering body surface area (BSA) of ≥3% and ≤10% and meet both of the following additional criteria:

   1. PASI score of ≥6 and ≤15, and
   2. PGA score of 2 or 3.

Key Exclusion Criteria:

1. Have a diagnosis of non-plaque psoriasis.
2. Plaque psoriasis restricted to scalp, palms, and soles only.
3. Have received systemic immunosuppressive therapy (MTX, apremilast, azathioprine, cyclosporine, 6-thioguanine, mercaptopurine, mycophenolate mofetil, hydroxyurea, and tacrolimus) within 4 weeks of first administration of study drug.
4. Unresponsive to prior use of biologics (including, but not limited to, TNFα inhibitors, natalizumab, efalizumab, anakinra or agents that modulate B cells or T cells).
5. If prior biologic therapy and responsive, participants must have been off therapy for at least 12 months prior to first administration of study drug.
6. Have received phototherapy or any systemic medications/treatments that could affect psoriasis or PGA evaluation (including, but not limited to oral or injectable corticosteroids, retinoids, psoralens, sulfasalazine, hydroxyurea, or fumaric acid derivatives) within 4 weeks of first administration of study drug. This includes therapeutic doses of non-steroidal anti-inflammatory drugs such as ibuprofen, although intermittent as required use as an analgesic is permitted when required. Chronic use of low dose aspirin for cardiovascular protection is permitted.
7. Currently receiving lithium, antimalarials, leflunomide, or IM gold, or have received lithium, antimalarials, IM gold, or leflunomide within 4 weeks of first administration of study drug.
8. Have used topical medications/treatments that could affect psoriasis or PGA evaluation (including [but not limited to] high- and mid-potency corticosteroids, anthralin, calcipotriene, topical vitamin D derivatives, retinoids, tazarotene, methoxsalen, trimethylpsoralens, picrolimus, and tacrolimus) within 2 weeks of the first administration of study drug. Topical unmedicated emollients and low-potency topical corticosteroids are not excluded.
9. Gastrointestinal tract disease (eg, short-bowel syndrome, diarrhea-predominant irritable bowel syndrome) that could interfere with GI delivery and transit time.
10. Active inflammatory bowel disease.
11. Active infection requiring systemic antiviral or antimicrobial therapy that will not be completed prior to Day 1 (Visit 2).
12. Have received live or live attenuated replicating vaccine within 6 weeks prior to screening or intend to have such a vaccination during the study.
13. Clinically significant abnormalities in screening laboratory values that would render a participant unsuitable for inclusion (per investigator judgment).
14. Known history of or positive test for HIV, or active infection with hepatitis C or chronic hepatitis B.
15. History of clinically significant acute cardiac or cerebrovascular event within 6 months before screening (includes stroke, transient ischemic attack, and coronary heart disease [angina pectoris, myocardial infarction, heart failure, revascularization procedures]).
16. Current acute or chronic inflammatory disease other than psoriasis or psoriatic arthritis (eg, inflammatory bowel disease, rheumatoid arthritis, systemic lupus erythematosus). If a subject is off all treatment and is disease and has been symptom free for greater than 12 months, then the inflammatory disease is considered to be in remission and they may be enrolled.
17. Hypersensitivity to P histicola or to any of the excipients.
18. Active untreated mental or psychiatric disorder. Participants who are on stable dosing of medication for a mental or psychiatric disorder for at least 6 months before screening and whose treating physicians consider them to be mentally stable may be enrolled.
19. Any major or minor GI surgery within 6 months of screening.
20. Any major surgery within 6 months of screening.
21. Malignancy within 5 years, except for basal or squamous cell carcinoma of the skin or carcinoma in situ of the cervix that has been successfully treated.
22. Treatment with another investigational drug, biological agent, or device within 1 month of screening, or 5 half-lives of investigational agent, whichever is longer.
23. Initiating any OTC or prescription medication including vitamins, herbal supplements and nutraceuticals (eg, supplements including high doses of probiotics and prebiotics as usually found in capsules/tablets/powders), except acetaminophen/paracetamol and anti-histamines, within 14 days prior to baseline or anticipates change in dosage for the duration of the study period. Note that probiotic and prebiotic foods that contain low doses are allowed (eg, yoghurt, kefir, kombucha, however, supplements containing high doses of probiotics and prebiotics are not allowed at any point during the study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 249 (Actual)
Dates: Start 2020-09-21 (Actual); Primary Completion 2021-07-02 (Actual); Study Completion 2021-12-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Ehst, MD PhD, Principal Investigator — Oregon Medical Research Center; Douglas Maslin, MPhil MBBS, Study Director — Evelo Biosciences
Locations (29):
- United States (8):
  - Synexus Clinical Research US, Inc. - Santa Rosa, Santa Rosa, California
  - Synexus Clinical Research US, Inc. - Orlando, Orlando, Florida
  - Synexus Clinical Research US, Inc. - St. Petersburg, St. Petersburg, Florida
  - ForCare Clinical Research, Tampa, Florida
  - Synexus Clinical Research US, Inc. - The Villages, The Villages, Florida
  - Synexus Clinical Research US, Inc. - Cincinnati, Cincinnati, Ohio
  - Oregon Medical Research Center PC, Portland, Oregon
  - Synexus Clinical Research US, Inc. - Anderson, Anderson, South Carolina
- Hungary (2):
  - Synexus Budapest - Magyarország Egészségügyi Szolgáltató Kft, Budapest
  - Synexus Zalaegerszeg Magyarország Egészségügyi Kft, Zalaegerszeg
- Poland (8):
  - Synexus - Poznan, Poznan, Greater Poland Voivodeship
  - Synexus - Wroclaw, Wroclaw, Lower Silesian Voivodeship
  - Synexus - Gdansk, Gdansk, Pomeranian Voivodeship
  - Synexus - Gdynia, Gdynia, Pomeranian Voivodeship
  - Synexus - Czestochowa, Częstochowa
  - Synexus - Katowice, Katowice
  - Synexus - Lodz, Lodz
  - Synexus - Warszawa, Warsaw
- United Kingdom (11):
  - Synexus - Thames Valley Clinical Research Centre, Reading, Berkshire
  - MAC Clinical Research, Blackpool, Lancashire
  - Synexus - Lancashire Clinical Research Centre, Chorley, Lancashire
  - Synexus - Merseyside Clinical Research Centre, Waterloo, Liverpool
  - Medicine Evaluation Unit, Wythenshawe, Manchester
  - MAC Clinical Research, Stockton-on-Tees, North Yorkshire
  - MAC Clinical Research, Cannock, Staffordshire
  - Synexus - Wales Clinical Research Centre, Cardiff, Wales
  - MAC Clinical Research, Leeds, West Yorkshire
  - Synexus - Scotland Clinical Research Centre, Glasgow
  - Synexus - Manchester Clinical Research Centre, Manchester

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ehst BD, Strober B, Blauvelt A, Maslin D, Macaro D, Carpenter N, Bodmer M, McHale D. A randomized, double-blinded, phase 2 trial of EDP1815, an oral immunomodulatory preparation of Prevotella histicola, in adults with mild-to-moderate plaque psoriasis. Front Med (Lausanne). 2024 May 15;11:1292406. doi: 10.3389/fmed.2024.1292406. eCollection 2024. PMID 38813388

RESULTS

PARTICIPANT FLOW:
Groups:
- Cohort 1 Active: 50 subjects with mild to moderate psoriasis on EDP1815 Dose = 0.8 x 10^11 cells, capsule, once daily, 16 weeks
- Cohort 1 Placebo: 25 subjects with mild to moderate psoriasis on placebo Dose = 0.8 x 10^11 cells, capsule, once daily, 16 weeks
- Cohort 2 Active: 50 subjects with mild to moderate psoriasis on EDP1815 Dose = 3.2 x 10^11 cells, capsule, once daily, 16 weeks
- Cohort 2 Placebo: 50 subjects with mild to moderate psoriasis on placebo Dose = 3.2 x 10^11 cells, capsule, once daily, 16 weeks
- Cohort 3 Active: 25 subjects with mild to moderate psoriasis on EDP1815 Dose = 8.0 x 10^11 cells, capsule, once daily, 16 weeks
- Cohort 3 Placebo: 25 subjects with mild to moderate psoriasis on placebo Dose = 8.0 x 10^11 cells, capsule, once daily, 16 weeks
Period: Overall Study
Arm/Group | Cohort 1 Active | Cohort 1 Placebo | Cohort 2 Active | Cohort 2 Placebo | Cohort 3 Active | Cohort 3 Placebo
Started | 56 | 28 | 55 | 27 | 55 | 28
Completed | 40 | 20 | 48 | 26 | 42 | 22
Not Completed | 16 | 8 | 7 | 1 | 13 | 6

BASELINE CHARACTERISTICS:
Groups:
- Cohort 1 Active: At least 50 subjects with mild to moderate psoriasis on EDP1815
  Dose = 0.8 x 10^11 cells, capsule, once daily, 16 weeks
- Cohort 1 Placebo: At least 25 subjects with mild to moderate psoriasis on placebo
  Dose = 0.8 x 10^11 cells, capsule, once daily, 16 weeks
- Cohort 2 Active: At least 50 subjects with mild to moderate psoriasis on EDP1815
  Dose = 3.2 x 10^11 cells, capsule, once daily, 16 weeks
- Cohort 2 Placebo: At least 25 subjects with mild to moderate psoriasis on placebo
  Dose = 3.2 x 10^11 cells, capsule, once daily, 16 weeks
- Cohort 3 Active: At least 50 subjects with mild to moderate psoriasis on EDP1815
  Dose = 8.0 x 10^11 cells, capsule, once daily, 16 weeks
- Cohort 3 Placebo: AT least 25 subjects with mild to moderate psoriasis on placebo.
  Dose = 8.0 x 10^11 cells, capsule, once daily, 16 weeks
- Total: Total of all reporting groups
Arm/Group | Cohort 1 Active | Cohort 1 Placebo | Cohort 2 Active | Cohort 2 Placebo | Cohort 3 Active | Cohort 3 Placebo | Total
Number analyzed (Participants) | 56 | 28 | 55 | 27 | 55 | 28 | 249
Age, Continuous [Median (Full Range); unit: years] | 44.0 [18 to 69] | 41.5 [22 to 64] | 42.0 [19 to 67] | 49.0 [23 to 68] | 44.0 [23 to 70] | 41.5 [19 to 64] | 43.0 [18 to 70]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 22 | 13 | 24 | 6 | 13 | 14 | 92
  Male | 34 | 15 | 31 | 21 | 42 | 14 | 157
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 1 | 1 | 1 | 0 | 1 | 7
  Not Hispanic or Latino | 53 | 27 | 54 | 26 | 55 | 26 | 241
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 1 | 1
Region of Enrollment [Number; unit: participants]
  Hungary | 3 | 1 | 5 | 1 | 2 | 1 | 13
  United States | 7 | 3 | 4 | 2 | 5 | 2 | 23
  Poland | 31 | 14 | 28 | 12 | 28 | 17 | 130
  United Kingdom | 15 | 10 | 18 | 12 | 20 | 8 | 83

OUTCOME MEASURES:

1. Primary Outcome: Mean Percentage Change in PASI
Description: The Psoriasis Area and Severity Index Score (PASI) is a physician assessment that combines the assessment of the severity of and area affected by psoriasis into a single score in the range 0 (no disease) to 72 (maximal disease).The efficacy of EDP1815 will be measured using the mean percentage change in PASI from baseline to week 16.
Time Frame: 16 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of change
Groups:
- All Placebo: 75 subjects with mild to moderate psoriasis on placebo, any dose
- Cohort 3 Active: 50 subjects with mild to moderate psoriasis on EDP1815
  Dose = 8.0 x 10^11 cells, capsule, once daily, 16 weeks
Arm/Group | All Placebo | Cohort 1 Active | Cohort 2 Active | Cohort 3 Active
Number analyzed (Participants) | 66 | 37 | 47 | 40
percentage of change | -14.39 [-22.66 to -5.52] | -20.37 [-31.65 to -9.47] | -22.73 [-33.08 to -11.88] | -23.49 [-34.18 to -12.12]
Statistical Analysis 1: Comparison: All Placebo vs Cohort 1 Active; Test type: Superiority; Posterior Mean difference = -5.99, 95% CI 2-sided [-20.28 to 7.12]
Statistical Analysis 2: Comparison: All Placebo vs Cohort 2 Active; Test type: Superiority; Posterior Mean difference = -8.35, 95% CI 2-sided [-22.07 to 5.04]
Statistical Analysis 3: Comparison: All Placebo vs Cohort 3 Active; Test type: Superiority; Posterior Mean difference = -9.10, 95% CI 2-sided [-23.22 to 4.65]

2. Secondary Outcome: Mean Percentage Change in PASI
Description: The Psoriasis Area and Severity Index Score (PASI) is a physician assessment that combines the assessment of the severity of and area affected by psoriasis into a single score in the range 0 (no disease) to 72 (maximal disease). The efficacy of EDP1815 will be measured using the mean percentage change from baseline in PASI from baseline at weeks 4, 8, and 12.
Time Frame: 12 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of change
Groups:
- All Placebo: 75 subjects with mild to moderate with psoriasis, on any dose
Arm/Group | All Placebo | Cohort 1 Active | Cohort 2 Active | Cohort 3 Active
Number analyzed (Participants) | 71 | 43 | 48 | 44
percentage of change | -19.24 [-26.17 to -11.57] | -21.84 [-31.85 to -12.91] | -22.57 [-31.32 to -13.05] | -19.13 [-28.77 to -9.83]
Statistical Analysis 1: Comparison: All Placebo vs Cohort 1 Active; Test type: Superiority; Posterior Mean difference = -2.60, 95% CI 2-sided [-13.91 to 9.90]
Statistical Analysis 2: Comparison: All Placebo vs Cohort 2 Active; Test type: Superiority; Posterior Mean difference = -3.33, 95% CI 2-sided [-15.21 to 8.52]
Statistical Analysis 3: Comparison: All Placebo vs Cohort 3 Active; Test type: Superiority; Posterior Mean difference = 0.11, 95% CI 2-sided [-12.33 to 11.53]

3. Secondary Outcome: Mean Absolute Change in PASI
Description: The Psoriasis Area and Severity Index Score (PASI) is a physician assessment that combines the assessment of the severity of and area affected by psoriasis into a single score in the range 0 (no disease) to 72 (maximal disease). The efficacy of EDP1815 will be measured using the mean absolute change from baseline in PASI from baseline at weeks 4, 8, 12, and 16.
Time Frame: 16 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | All Placebo | Cohort 1 Active | Cohort 2 Active | Cohort 3 Active
Number analyzed (Participants) | 66 | 37 | 47 | 40
score on a scale | -1.16 [-1.87 to -0.41] | -1.85 [-2.74 to -0.91] | -1.88 [-2.77 to -1.04] | -1.97 [-2.92 to -1.08]
Statistical Analysis 1: Comparison: All Placebo vs Cohort 1 Active; Test type: Superiority; Posterior Mean difference = -0.69, 95% CI 2-sided [-1.88 to 0.46]
Statistical Analysis 2: Comparison: All Placebo vs Cohort 2 Active; Test type: Superiority; Posterior Mean difference = -0.73, 95% CI 2-sided [-1.82 to 0.45]
Statistical Analysis 3: Comparison: All Placebo vs Cohort 3 Active; Test type: Superiority; Posterior Mean difference = -0.81, 95% CI 2-sided [-2.05 to 0.33]

4. Secondary Outcome: Achievement of PASI-50
Description: The efficacy of EDP1815 will be measured using the achievement of PASI-50 at weeks 4, 8, 12, and 16. PASI-50 is defined by at least a 50% reduction from baseline in the PASI score.
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | All Placebo | Cohort 1 Active | Cohort 2 Active | Cohort 3 Active
Number analyzed (Participants) | 66 | 37 | 47 | 40
Participants | 8 | 11 | 15 | 10
Statistical Analysis 1: Comparison: All Placebo vs Cohort 3 Active; Test type: Superiority; Odds Ratio (OR) = 2.64, 95% CI 2-sided [1.01 to 6.94]
Statistical Analysis 2: Comparison: All Placebo vs Cohort 2 Active; Test type: Superiority; Odds Ratio (OR) = 2.93, 95% CI 2-sided [1.17 to 7.37]
Statistical Analysis 3: Comparison: All Placebo vs Cohort 3 Active; Test type: Superiority; Odds Ratio (OR) = 1.73, 95% CI 2-sided [0.63 to 4.70]

5. Secondary Outcome: Time to First Achievement of PASI-50
Description: The efficacy of EDP1815 will be measured using the time to first achievement of PASI-50
Time Frame: 20 weeks
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | All Placebo | Cohort 1 Active | Cohort 2 Active | Cohort 3 Active
Number analyzed (Participants) | 83 | 56 | 55 | 55
days | 160 [160 to NA] — Insufficient number of participants with event. | NA [NA to NA] — Insufficient number of participants with event. | NA [NA to NA] — Insufficient number of participants with event. | 146 [146 to 154]
Statistical Analysis 1: Comparison: All Placebo vs Cohort 1 Active; Test type: Superiority; p = 0.100, nonparametric survival analysis; Method used was a nonparametric survival analysis for interval censored data
Statistical Analysis 2: Comparison: All Placebo vs Cohort 2 Active; Test type: Superiority; p = 0.034, nonparametric survival analysis; Method used was a nonparametric survival analysis for interval censored data
Statistical Analysis 3: Comparison: All Placebo vs Cohort 3 Active; Test type: Superiority; p = 0.094, nonparametric survival analysis; Method used was a nonparametric survival analysis for interval censored data

6. Secondary Outcome: Achievement of PASI-75
Description: The efficacy of EDP1815 will be measured using the achievement of PASI-75 at week 16. PASI-75 response is defined by at least a 75% reduction from baseline in the PASI score.
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | All Placebo | Cohort 1 Active | Cohort 2 Active | Cohort 3 Active
Number analyzed (Participants) | 66 | 37 | 47 | 40
Participants | 2 | 2 | 4 | 4

7. Secondary Outcome: Achievement of PASI-90
Description: The efficacy of EDP1815 will be measured using the achievement of PASI-90 at week 16.PASI-90 response is defined by at least a 90% reduction from baseline in the PASI score.
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | All Placebo | Cohort 1 Active | Cohort 2 Active | Cohort 3 Active
Number analyzed (Participants) | 66 | 37 | 47 | 40
Participants | 0 | 2 | 2 | 0

8. Secondary Outcome: Achievement of PASI-100
Description: The efficacy of EDP1815 will be measured using the achievement of PASI-100 at week 16. PASI-100 response is defined as achieving a complete resolution of all disease.
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | All Placebo | Cohort 1 Active | Cohort 2 Active | Cohort 3 Active
Number analyzed (Participants) | 66 | 37 | 47 | 40
Participants | 0 | 0 | 0 | 0

9. Secondary Outcome: Achievement of PGA of 0 or 1 With a ≥2-point Improvement From Baseline
Description: The efficacy of EDP1815 will be measured using the achievement of PGA of 0 or 1 with a ≥2-point improvement from baseline at Week 16 [PGA = Physician's Global Assessment]. The National Psoriasis Foundation Psoriasis Score version of a PGA is calculated by averaging the total body erythema, induration, and desquamation scores. Erythema, induration, and desquamation will be scored on a 6-point scale, ranging from 0 (clear) to 5 (severe): the total PGA score is defined as the average of the erythema, induration, and desquamation scores. PGA score of 0 or 1 is defined as clear or almost clear of psoriasis.
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | All Placebo | Cohort 1 Active | Cohort 2 Active | Cohort 3 Active
Number analyzed (Participants) | 66 | 37 | 47 | 40
Participants | 4 | 4 | 5 | 5
Statistical Analysis 1: Comparison: All Placebo vs Cohort 1 Active; Test type: Superiority; Posterior Mean Odds Ratio = 2.14, 95% CI 2-sided [0.45 to 10.96]
Statistical Analysis 2: Comparison: All Placebo vs Cohort 2 Active; Test type: Superiority; Posterior Mean Odds Ratio = 2.02, 95% CI 2-sided [0.42 to 8.78]
Statistical Analysis 3: Comparison: All Placebo vs Cohort 3 Active; Test type: Superiority; Posterior Mean Odds Ratio = 2.12, 95% CI 2-sided [0.46 to 9.51]

10. Secondary Outcome: Achievement of PGA of 0
Description: The efficacy of EDP1815 will be measured using the achievement of PGA of 0 at Week 16 [PGA = Physician's Global Assessment]. The National Psoriasis Foundation Psoriasis Score version of a PGA is calculated by averaging the total body erythema, induration, and desquamation scores. Erythema, induration, and desquamation will be scored on a 6-point scale, ranging from 0 (clear) to 5 (severe): the total PGA score is defined as the average of the erythema, induration, and desquamation scores. PGA score of 0 or 1 is defined as clear or almost clear of psoriasis. A PGA 0 is defined as clear or no signs of psoriasis.
Time Frame: 16 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | All Placebo | Cohort 1 Active | Cohort 2 Active | Cohort 3 Active
Number analyzed (Participants) | 66 | 37 | 47 | 40
Participants | 1 | 0 | 0 | 1
Statistical Analysis 1: Comparison: All Placebo vs Cohort 1 Active; Test type: Superiority; There were not enough responders to model using GLMM or a Bayesian logistic model, and no treatment difference analysis was conducted
Statistical Analysis 2: Comparison: All Placebo vs Cohort 2 Active; Test type: Superiority; [other analysis details as in outcome 10, analysis 1]
Statistical Analysis 3: Comparison: All Placebo vs Cohort 3 Active; Test type: Superiority; [other analysis details as in outcome 10, analysis 1]

11. Secondary Outcome: Mean Percentage Change in PGAxBSA
Description: [PGA = Physician's Global Assessment, BSA = Body Surface Area]. The National Psoriasis Foundation Psoriasis Score version of a static Physicians Global Asessment (PGA) is calculated by averaging the total body erythema, induration, and desquamation scores. Erythema, induration, and desquamation will be scored on a 6-point scale, ranging from 0 (clear) to 5 (severe): the total PGA score is defined as the average of the erythema, induration, and desquamation scores.
  Body surface area (BSA) measures the total area of the body affected by psoriasis. Psoriasis that occurs on less than 5 percent of the BSA is considered mild to moderate psoriasis. Psoriasis affecting more than 5 percent of the BSA is considered moderate to severe psoriasis.
  The efficacy of EDP1815 will be measured using the mean percentage change from baseline in PGA x BSA at Weeks 4, 8, 12, and 16.
Time Frame: 16 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of change
Arm/Group | All Placebo | Cohort 1 Active | Cohort 2 Active | Cohort 3 Active
Number analyzed (Participants) | 66 | 37 | 47 | 40
percentage of change | -0.05 [-13.65 to 12.74] | -9.13 [-25.84 to 7.91] | -3.04 [-19.15 to 12.26] | -17.16 [-33.23 to -1.18]
Statistical Analysis 1: Comparison: All Placebo vs Cohort 1 Active; Test type: Superiority; Posterior Mean difference = -9.08, 95% CI 2-sided [-30.22 to 12.40]
Statistical Analysis 2: Comparison: All Placebo vs Cohort 2 Active; Test type: Superiority; Posterior Mean difference = 2.99, 95% CI 2-sided [-23.41 to 18.15]
Statistical Analysis 3: Comparison: All Placebo vs Cohort 3 Active; Test type: Superiority; Posterior Mean difference = -17.10, 95% CI 2-sided [-38.29 to 3.25]

12. Secondary Outcome: Mean Absolute Change in PGAxBSA
Description: [PGA = Physician's Global Assessment, BSA = Body Surface Area]. The National Psoriasis Foundation Psoriasis Score version of a static Physicians Global Asessment (PGA) is calculated by averaging the total body erythema, induration, and desquamation scores. Erythema, induration, and desquamation will be scored on a 6-point scale, ranging from 0 (clear) to 5 (severe): the total PGA score is defined as the average of the erythema, induration, and desquamation scores.
  Body surface area (BSA) measures the total area of the body affected by psoriasis. Psoriasis that occurs on less than 5 percent of the BSA is considered mild to moderate psoriasis. Psoriasis affecting more than 5 percent of the BSA is considered moderate to severe psoriasis.
  The efficacy of EDP1815 will be measured using the mean absolute change from baseline in PGA x BSA at Weeks 4, 8, 12, and 16.
Time Frame: 16 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | All Placebo | Cohort 1 Active | Cohort 2 Active | Cohort 3 Active
Number analyzed (Participants) | 66 | 37 | 47 | 40
score on a scale | -0.01 [-2.68 to 2.41] | -2.67 [-5.77 to 0.60] | -0.84 [-3.93 to 2.06] | -3.54 [-6.58 to -0.29]
Statistical Analysis 1: Comparison: All Placebo vs Cohort 1 Active; Test type: Superiority; Posterior Mean difference = -2.66, 95% CI 2-sided [-6.79 to 1.52]
Statistical Analysis 2: Comparison: All Placebo vs Cohort 2 Active; Test type: Superiority; Posterior Mean difference = -0.83, 95% CI 2-sided [-4.70 to 3.16]
Statistical Analysis 3: Comparison: All Placebo vs Cohort 3 Active; Test type: Superiority; Posterior Mean difference = -3.53, 95% CI 2-sided [-7.49 to 0.63]

13. Secondary Outcome: Mean Percentage Change in LSS
Description: The LSS is used to score the severity of psoriasis plaques. The dimensions of scaling, erythema, and plaque elevation are each scored on a scale from 0 (clear) to 4 (very severe), and the total LSS is the numerical sum of the 3-dimensional scores. The efficacy of EDP1815 will be measured using the mean percentage change from baseline in LSS (Lesion Severity Score) at Weeks 4, 8, 12, and 16.
Time Frame: 16 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of change
Arm/Group | All Placebo | Cohort 1 Active | Cohort 2 Active | Cohort 3 Active
Number analyzed (Participants) | 66 | 36 | 46 | 39
percentage of change | -14.11 [-22.19 to -5.99] | -21.06 [-31.72 to -10.02] | -16.46 [-26.62 to -6.82] | -16.16 [-26.65 to -5.18]
Statistical Analysis 1: Comparison: All Placebo vs Cohort 1 Active; Test type: Superiority; Posterior Mean difference = -9.08, 95% CI 2-sided [-30.22 to 12.40]
Statistical Analysis 2: Comparison: All Placebo vs Cohort 2 Active; Test type: Superiority; Posterior Mean difference = -2.99, 95% CI 2-sided [-23.41 to 18.15]
Statistical Analysis 3: Comparison: All Placebo vs Cohort 3 Active; Test type: Superiority; Posterior Mean difference = -17.10, 95% CI 2-sided [-38.29 to 3.25]

14. Secondary Outcome: Mean Absolute Change in LSS
Description: The LSS is used to score the severity of psoriasis plaques. The dimensions of scaling, erythema, and plaque elevation are each scored on a scale from 0 (clear) to 4 (very severe), and the total LSS is the numerical sum of the 3-dimensional scores.The efficacy of EDP1815 will be measured using the mean absolute change from baseline in LSS (Lesion Severity Score) at Weeks 4, 8, 12, and 16.
Time Frame: 16 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | All Placebo | Cohort 1 Active | Cohort 2 Active | Cohort 3 Active
Number analyzed (Participants) | 66 | 36 | 46 | 39
score on a scale | -1.13 [-1.62 to -0.67] | -1.37 [-1.97 to -0.71] | -1.08 [-1.70 to -0.49] | -1.03 [-1.66 to -0.40]
Statistical Analysis 1: Comparison: All Placebo vs Cohort 1 Active; Test type: Superiority; Posterior Mean difference = -2.66, 95% CI 2-sided [-6.79 to 1.52]
Statistical Analysis 2: Comparison: All Placebo vs Cohort 2 Active; Test type: Superiority; Posterior Mean difference = -0.83, 95% CI 2-sided [-4.70 to 3.16]
Statistical Analysis 3: Comparison: All Placebo vs Cohort 3 Active; Test type: Superiority; Posterior Mean difference = -3.53, 95% CI 2-sided [-7.49 to 0.63]

15. Secondary Outcome: Mean Percentage Change in DLQI
Description: The DLQI is a patient reported outcomes instrument for assessing the impact of dermatologic conditions on patients' quality of life. The higher the score the more the impact on quality of life. The efficacy of EDP1815 will be measured using mean percentage change from baseline in Dermatology Life Quality Index (DLQI) at Weeks 4, 8, 12, and 16.
Time Frame: 16 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of change
Arm/Group | All Placebo | Cohort 1 Active | Cohort 2 Active | Cohort 3 Active
Number analyzed (Participants) | 64 | 37 | 47 | 40
percentage of change | -26.45 [-41.20 to -10.72] | -23.46 [-42.34 to -4.39] | -28.94 [-46.16 to -9.79] | -13.09 [-32.20 to 5.38]
Statistical Analysis 1: Comparison: All Placebo vs Cohort 1 Active; Test type: Superiority; Posterior Mean difference = 2.99, 95% CI 2-sided [-19.99 to 28.84]
Statistical Analysis 2: Comparison: All Placebo vs Cohort 2 Active; Test type: Superiority; Posterior Mean difference = -2.49, 95% CI 2-sided [-26.47 to 21.55]
Statistical Analysis 3: Comparison: All Placebo vs Cohort 3 Active; Test type: Superiority; Posterior Mean difference = 13.36, 95% CI 2-sided [-12.03 to 36.92]

16. Secondary Outcome: Mean Absolute Change in DLQI
Description: The DLQI is a patient reported outcomes instrument for assessing the impact of dermatologic conditions on patients' quality of life. There are 10 questions each scored 0-3, the higher the score the more the impact on quality of life (Total score range 0-30; 0 = no impact, 30 = greatest impact).The efficacy of EDP1815 will be measured using the mean absolute change from baseline in Dermatology Life Quality Index (DLQI) at Weeks 4, 8, 12, and 16
Time Frame: 16 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | All Placebo | Cohort 1 Active | Cohort 2 Active | Cohort 3 Active
Number analyzed (Participants) | 66 | 37 | 47 | 40
score on a scale | -2.42 [-3.50 to -1.38] | -1.80 [-3.19 to -0.51] | -2.63 [-3.90 to -1.38] | -2.50 [-3.91 to -1.18]
Statistical Analysis 1: Comparison: All Placebo vs Cohort 1 Active; Test type: Superiority; Posterior Mean difference = 0.62, 95% CI 2-sided [-1.10 to 2.30]
Statistical Analysis 2: Comparison: All Placebo vs Cohort 2 Active; Test type: Superiority; Posterior Mean difference = -0.21, 95% CI 2-sided [-1.96 to 1.37]
Statistical Analysis 3: Comparison: All Placebo vs Cohort 3 Active; Test type: Superiority; Posterior Mean difference = -0.08, 95% CI 2-sided [-1.73 to 1.75]

17. Secondary Outcome: Mean Percentage Change in mNAPSI
Description: The mNAPSI is a tool for physicians to evaluate the severity of nail bed psoriasis and nail matrix psoriasis by area of involvement in the nail unit. The higher the score the more severe the nail bed psoriasis. The efficacy of EDP1815 will be measured using the mean percentage change in mNAPSI total score (modified Nail Psoriasis Severity Index) from baseline at Weeks 4, 8, 12, and 16
Time Frame: 16 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: percentage of change
Arm/Group | All Placebo | Cohort 1 Active | Cohort 2 Active | Cohort 3 Active
Number analyzed (Participants) | 35 | 12 | 23 | 25
percentage of change | -5.28 [-35.93 to 29.58] | 8.43 [-44.63 to 60.13] | 68.41 [25.97 to 109.34] | 3.13 [-37.13 to 41.16]
Statistical Analysis 1: Comparison: All Placebo vs Cohort 1 Active; Test type: Superiority; Posterior Mean difference = 13.71, 95% CI 2-sided [-50.62 to 73.35]
Statistical Analysis 2: Comparison: All Placebo vs Cohort 2 Active; Test type: Superiority; Posterior Mean difference = 73.69, 95% CI 2-sided [21.69 to 126.92]
Statistical Analysis 3: Comparison: All Placebo vs Cohort 3 Active; Test type: Superiority; Posterior Mean difference = 8.41, 95% CI 2-sided [-44.58 to 56.81]

18. Secondary Outcome: Mean Absolute Change in mNAPSI
Description: The mNAPSI is a tool for physicians to evaluate the severity of nail bed psoriasis and nail matrix psoriasis by area of involvement in the nail unit. Each fingernail is rated for the presence and severity of seven features to give a total fingernail score of 0-13 (0= no involvement, 13 = greatest involvement). The total mNAPSI score is the sum of the 10 fingernail scores (range 0-130; 0= no involvement, 130= greatest involvement).The higher the score the more severe the nail bed psoriasis. The efficacy of EDP1815 will be measured using the mean absolute change in mNAPSI total score (modified Nail Psoriasis Severity Index) from baseline at Weeks 4, 8, 12, and 16
Time Frame: 16 weeks
Measure: Least Squares Mean (95% Confidence Interval); unit: score on a scale
Arm/Group | All Placebo | Cohort 1 Active | Cohort 2 Active | Cohort 3 Active
Number analyzed (Participants) | 35 | 12 | 23 | 25
score on a scale | -1.22 [-4.70 to 2.33] | -0.97 [-6.44 to 4.89] | 1.13 [-3.43 to 5.65] | -0.14 [-4.47 to 3.99]
Statistical Analysis 1: Comparison: All Placebo vs Cohort 1 Active; Test type: Superiority; Posterior Mean difference = 0.62, 95% CI 2-sided [-1.10 to 2.30]
Statistical Analysis 2: Comparison: All Placebo vs Cohort 2 Active; Test type: Superiority; Posterior Mean difference = -0.21, 95% CI 2-sided [-1.96 to 1.37]
Statistical Analysis 3: Comparison: All Placebo vs Cohort 3 Active; Test type: Superiority; Posterior Mean difference = -0.08, 95% CI 2-sided [-1.73 to 1.75]

19. Secondary Outcome: Cumulative Incidence of Partial Relapse
Description: The efficacy of EDP1815 will be measured by calculating the cumulative incidence of partial relapse at Weeks 20, 24, 28, and 40 for participants who were classified as responders at week 16. Partial relapse is defined as a loss of the PASI-50 response after week 16 and after cessation of study treatment, or commencing a new treatment for psoriasis.
Time Frame: 40 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | All Placebo | Cohort 1 Active | Cohort 2 Active | Cohort 3 Active
Number analyzed (Participants) | 9 | 12 | 16 | 10
Participants | 4 | 4 | 8 | 2

20. Secondary Outcome: Cumulative Incidence of Complete Relapse
Description: The efficacy of EDP1815 will be measured by calculating the cumulative incidence of complete relapse at Weeks 20, 24, 28, and 40 in participants who were considered as responders at week 16. Relapse is defined as an increase in the severity of the psoriasis as measured by PASI to the baseline value or greater, or commencement of a new treatment for psoriasis.
Time Frame: 40 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | All Placebo | Cohort 1 Active | Cohort 2 Active | Cohort 3 Active
Number analyzed (Participants) | 9 | 12 | 16 | 10
Participants | 0 | 1 | 2 | 1

21. Secondary Outcome: Cumulative Incidence of Rebound
Description: The efficacy of EDP1815 will be measured by calculating the cumulative incidence of rebound at Weeks 20, 24, 28, and 40 in participants with at least one PASI assessment after the end of treatment. Rebound is defined as an increase in the severity of the psoriasis as measured by PASI to 125% of baseline score or above, or onset of new pustular/erythrodermic psoriasis, within 3 months of cessation of study treatment.
Time Frame: 40 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | All Placebo | Cohort 1 Active | Cohort 2 Active | Cohort 3 Active
Number analyzed (Participants) | 64 | 37 | 43 | 45
Participants | 7 | 6 | 3 | 1

ADVERSE EVENTS:
Time Frame: Adverse event (AE) data were collected over a period of 20 weeks.
Arm/Group | All Placebo | Cohort 1 Active | Cohort 2 Active | Cohort 3 Active
All-Cause Mortality (participants affected / at risk) | 0/83 | 0/56 | 0/55 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/83 | 1/56 | 0/55 | 1/55
Other Adverse Events (participants affected / at risk) | 22/83 | 21/56 | 21/55 | 25/55
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Placebo (N=83) | Cohort 1 Active (N=56) | Cohort 2 Active (N=55) | Cohort 3 Active (N=55)
COVID-19 Pneumonia (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Peptic Ulcer Hemorrhage (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | All Placebo (N=83) | Cohort 1 Active (N=56) | Cohort 2 Active (N=55) | Cohort 3 Active (N=55)
COVID-19 (Infections and infestations) | 4 (4) | 2 (2) | 3 (3) | 1 (1)
Viral Upper Respiratory Tract Infection (Infections and infestations) | 0 (0) | 2 (2) | 3 (3) | 1 (1)
Upper Respiratory Tract Infection (Infections and infestations) | 1 (1) | 4 (5) | 0 (0) | 5 (6)
Headache (Nervous system disorders) | 9 (15) | 7 (20) | 3 (5) | 5 (8)
Diarrhea (Gastrointestinal disorders) | 5 (6) | 2 (2) | 1 (1) | 4 (6)
Abdominal Pain (Gastrointestinal disorders) | 2 (2) | 1 (2) | 3 (4) | 2 (2)
Dyspepsia (Gastrointestinal disorders) | 2 (2) | 0 (0) | 4 (7) | 2 (2)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 3 (3) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 3 (3)
Vaccination Complication (Injury, poisoning and procedural complications) | 3 (3) | 2 (2) | 1 (1) | 5 (5)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
After completion of the study, the data may be considered for reporting at a scientific meeting or for publication in a scientific journal. The sponsor has final approval authority over publication of the study data.

DOCUMENTS (2):
  • Study Protocol (2020-11-17): https://cdn.clinicaltrials.gov/large-docs/27/NCT04603027/Prot_000.pdf
  • Statistical Analysis Plan (2021-07-23): https://cdn.clinicaltrials.gov/large-docs/27/NCT04603027/SAP_001.pdf